CLINICAL TRIAL: NCT06550531
Title: Impact of Human Papillomavirus Carriage on IVF/ICSI Results at Brest University Hospital
Brief Title: Impact of Human Papillomavirus Carriage on IVF/ICSI Results (HPV AMP)
Acronym: HPV-AMP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0363 - HPV AMP
Record Dates: First submitted 2022-03-31; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Human Papilloma Virus; Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The prevalence of the papilloma virus in the general population is 12%. This virus is known to impair male fertility but its impact on female infertility remains uncertain. This is a public health problem since there is a vaccination protocol. Demonstrating the impact of the human papillomavirus on fertility would be an argument in favor of vaccination.

DETAILED DESCRIPTION:
This is a single-center prospective study in the assisted reproduction center of Brest University Hospital. All new patients coming to consult will be offered participation in the study. The HPV test will be updated if it is older than 12 months. We will analyze stimulation results and pregnancy outcomes according to HPV status. Inclusions will take place over 3 years

ELIGIBILITY:
Inclusion Criteria:

* all etiology of infertility AMH > ou = à 1.1 ng/ml First ou second protocol of IVF between 25 years and 37 years and 11 months

Exclusion Criteria:

Age < 25 y Age > ou = 38 y AMH < 1.1 ng/ml patient under juridic protection rejection of participation

Ages: 25 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population study is a population of infertile women who are consulting in our center of Reproduction Médicine in CHU Brest.
Sampling Method: Non-Probability Sample
Enrollment: 618 (Estimated)
Dates: Start 2022-02-04 (Actual); Primary Completion 2026-02-04 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate after fresh eSET by HPV status | 1 year
  A clinical pregancy is the visualisation of a gestational sac inside the uterus after 6 weeks of gestation

SECONDARY OUTCOMES:
IVF issues | 1 year
  oocytes number, embryos number, fecondation rate, implantation rate
Positive HPV rate | 1 year
  number of women who have a positive HPV test before IVF procedure

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning four years and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.